CLINICAL TRIAL: NCT02410928
Title: Comparison of the Vocal Cord Imaging Techniques After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, DR, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: USG-Vokal cord
Record Dates: First submitted 2015-02-14; First posted 2015-04-08 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2015-02

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fiberoptic nasal laringoscopy (Experimental): the vocal cords ill be visualized with fiberoptic nasal laringoscopy
  Interventions: Device: fiberoptic nasal laringoscopy
- ultrasonography (Experimental): the vocal cords ill be visualized with ultrasonography
  Interventions: Device: ultrasonograph
- Direct laringoscopy (Active Comparator): the vocal cords ill be visualized with direct laringoscopy
  Interventions: Device: direct laringoscopy

INTERVENTIONS:
Device: direct laringoscopy — the vocal cords will be visualized after extubation with direct laringoscopy
  Other Names: direct laryngoscopy
  Arms: Direct laringoscopy
Device: fiberoptic nasal laringoscopy — the vocal cords will be visualized after extubation with fiberoptic nasal laringoscopy
  Other Names: fiberoptic laryngoscopy
  Arms: fiberoptic nasal laringoscopy
Device: ultrasonograph — the vocal cords will be visualized after extubation with fiberoptic ultrasonography
  Other Names: ultrsonography
  Arms: ultrasonography

SUMMARY:
Recurrent nerve palsy is a complication of thyroidectomy. Most surgeons want to visualize the vocal cords after tyroidectomy. The aim is to compare the direct laringoscopy, videolaringoscopy, fiberoptic laringoscopy and ultrasonography methods in terms of efficacy, duration and hemodynamic responses during the procedure.

DETAILED DESCRIPTION:
The vocal cord will be visualised after the extubation with one of the following methods:

direct laringoscopy videolaringoscopy fiberoptic laringoscopy ultrasonography The of efficacy of the method (0= not able to visualize the vocal cords, 1= the vocal cords were visualized) duration of the procedure and hemodynamic responses (heart rate, mean arterial pressure) during the procedure will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Benign or malignant thyroid pathology

Exclusion Criteria:

* anticipated difficult intubation

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
visualisation of the vocal cords | 1 min after extubation
  the vocal cords will be examined after extubation
duration of the procedure | 10 min after extubation
  the duration of the vocal cord examination
mean arterial pressure | 10 min after extubation
  the mean arterial pressure will be measured after extubation
heart rate | 10 min after extubation
  the heart rate will be measured after extubation
peripheal oxygen saturation | 10 min after extubation
  the peripheal oxygen saturation will be measured after extubation

SECONDARY OUTCOMES:
hypertention | 5 minutes after the extubation
  mean arterial pressure >20% from baseline value
tachycardia | 5 minutes after the extubation
  heart rate >20% from baseline value
laceration | 5 minutes after the extubation
  blood detected on the blade/fiber optic scope, or macroscopic blood on the oral nasal mucosa
teeht damage | 5 minutes after the extubation
  broken teeht

CONTACTS AND LOCATIONS:
Overall Officials: Dilek yazicioglu, Dr, Study Director — Diskapi Teaching and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Jeannon JP, Orabi AA, Bruch GA, Abdalsalam HA, Simo R. Diagnosis of recurrent laryngeal nerve palsy after thyroidectomy: a systematic review. Int J Clin Pract. 2009 Apr;63(4):624-9. doi: 10.1111/j.1742-1241.2008.01875.x. PMID 19335706
- [Result] Higgins TS, Gupta R, Ketcham AS, Sataloff RT, Wadsworth JT, Sinacori JT. Recurrent laryngeal nerve monitoring versus identification alone on post-thyroidectomy true vocal fold palsy: a meta-analysis. Laryngoscope. 2011 May;121(5):1009-17. doi: 10.1002/lary.21578. PMID 21520117
- [Result] Kristensen MS. Ultrasonography in the management of the airway. Acta Anaesthesiol Scand. 2011 Nov;55(10):1155-73. doi: 10.1111/j.1399-6576.2011.02518.x. Epub 2011 Sep 7. PMID 22092121